CLINICAL TRIAL: NCT03104231
Title: OCULUS: a 3-D Movie to Improve Patient Compliance
Brief Title: VR-3D Movie-based Education
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of Warsaw (Other)
Responsible Party: Principal Investigator, Marcin Grabowski, Ass. Prof, Medical University of Warsaw
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: OCULUS
Record Dates: First submitted 2017-03-28; First posted 2017-04-07 (Actual); Last update posted 2017-06-08 (Actual); Status verified 2017-06

CONDITIONS: mHealth
Keywords: atrial fibrillation; oral anticoagulantion; stroke prevention; education; e-medicine
MeSH Terms: conditions — Atrial Fibrillation | interventions — Motion Pictures

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- study group (Experimental): All the patients will be shown three-dimensional (3D) movie.
  Interventions: Other: three-dimensional (3D) movie

INTERVENTIONS:
Other: three-dimensional (3D) movie — Brief VR-3D will be shown using the oculus glasses and a smartphone. Then, patients will be asked several questions from the prepared questionnaire.

SUMMARY:
Atrial fibrillation (AF), which is the most common cardiac arrhythmia in adults, is associated with a high risk of stroke and other thromboembolic complications. The usage of oral anticoagulation (OAC) may prevent the incidence of the thromboembolic events in the majority of patients. The current guidelines for the management of AF patients highlight the important role of patients' education, since the clinical benefit from OAC treatment may be achieved by the effective cooperation between patients and physicians. It has been suggested, that compliance may be increased by the novel e-solutions introduced into the daily clinical practice. Due to the improvement in advanced technologies, the virtual reality (VR) three-dimensional (3D) movie stands for a future alternative in e-medicine. The aim of the OCULUS study was to examine whether the 3D movie-based knowledge transfer is effective in teaching patients about the consequences of AF and pharmacological possibilities in reducing the risk of stroke.

DETAILED DESCRIPTION:
The OCULUS is a prospective, single centre study. The study will include hospitalized patients, who are over 18 years old. The only exclusion criteria of the study is the previously diagnosed dementia. The study is based on the questionnaire designed by the authors of the study, enclosing questions about sex, age, education, current job, AF history and knowledge about consequences of AF and the possibility of stroke prevention due to the OAC therapy. Subsequently, the brief VR-3D will be shown using the oculus glasses and a smartphone. The movie's plot informs about the risk of stroke and importance of the OAC therapy to prevent the incidence of the thromboembolic complications of AF. Consequently, patients will be asked several questions, including what was the movie about, whether AF can affect patient's life in a negative way, is it possible to reduce the risk of stroke and by what kind of drugs. Similar questions will be asked to the patients immediately after the movie, one week and one year later, via the Telephone follow-up.

ELIGIBILITY:
Inclusion Criteria:

* >18 years old
* signed written informed consent

Exclusion Criteria:

* previously diagnosed dementia

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2016-04-01 (Actual); Primary Completion 2017-04-30 (Actual); Study Completion 2017-05-30 (Actual)

PRIMARY OUTCOMES:
Assessment of the effectiveness of the 3D-movie based knowledge transfer in teaching patients about the consequences of AF | 1 year
  The outcome will be assessed by questionnaire designed by the authors of the study, enclosing questions about sex, age, education, current job, AF history and knowledge about consequences of AF and the possibility of stroke prevention due to the OAC therapy.

CONTACTS AND LOCATIONS:
Overall Officials: Paweł Balsam, MD, PhD, Principal Investigator — 1st Chair and Department of Cardiology, Medical University of Warsaw, Warsaw, Poland
Locations (1):
- Paweł Balsam, Warsaw, Poland

IPD SHARING:
Plan to Share IPD: Yes
We will be able to share all of the data. They will be available on april 2017th.

REFERENCES:
- [Derived] Balsam P, Borodzicz S, Malesa K, Puchta D, Tyminska A, Ozieranski K, Koltowski L, Peller M, Grabowski M, Filipiak KJ, Opolski G. OCULUS study: Virtual reality-based education in daily clinical practice. Cardiol J. 2019;26(3):260-264. doi: 10.5603/CJ.a2017.0154. Epub 2018 Jan 3. PMID 29297178